CLINICAL TRIAL: NCT05344040
Title: Remote Exercise Effects on Cognitive Processing Speed in Multiple Sclerosis: A Pilot Trial
Acronym: REACT-MS
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Kessler Foundation (Other)
Responsible Party: Principal Investigator, Brian Sandroff, Principal Investigator, Kessler Foundation
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E-1197-22
Record Dates: First submitted 2022-04-13; First posted 2022-04-25 (Actual); Last update posted 2022-12-05 (Actual); Status verified 2022-12

CONDITIONS: Multiple Sclerosis
Keywords: Exercise; Physical Activity; Cognition; Walking; Stretching
MeSH Terms: conditions — Multiple Sclerosis; Motor Activity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Remotely Delivered and Supported Aerobic Walking Exercise Training (Experimental)
  Interventions: Behavioral: Remotely Delivered and Supported Aerobic Walking Exercise Training
- Remotely Delivered and Supported Stretching and Toning (Active Comparator)
  Interventions: Behavioral: Remotely Delivered and Supported Stretching and Toning Exercise Training

INTERVENTIONS:
Behavioral: Remotely Delivered and Supported Aerobic Walking Exercise Training — This condition will include 16-weeks of remotely-delivered and supported aerobic walking exercise training based on guidelines for physical activity in persons with MS for general health benefits. Exercise intensities will be prescribed based on steps per exercise sessions from a waist-worn FitBit One™ (FitBit, Inc., San Francisco, CA).
  The exercise program involves one-on-one semi-structured sessions with an MS exercise specialist (i.e., behavior coach) throughout the program. These sessions focus on exercise training guidance and oversight, discussion of the behavioral strategies of action planning and self-monitoring, and presentation and discussion of newsletters for optimizing exercise compliance.
  Arms: Remotely Delivered and Supported Aerobic Walking Exercise Training
Behavioral: Remotely Delivered and Supported Stretching and Toning Exercise Training — The active, non-aerobic exercise condition will involve stretching-and-toning activities. These activities will be based on a manual provided by the National Multiple Sclerosis Society. Participants will be provided with necessary exercise equipment (e.g., yoga mat, FitBit), an instructional DVD, and a manual, log-book, calendar, and prescription for the stretching program. This program will be supplemented with periodic newsletters delivered electronically that highlight principles of behavior change, and video-chats with a behavior coach that provide motivation and social accountability. These occur on the same timeline and frequency as in the walking condition, but focus on constructs for stretching.
  Arms: Remotely Delivered and Supported Stretching and Toning

SUMMARY:
Cognitive processing speed (CPS) impairment is prevalent, impactful, and poorly-managed in multiple sclerosis (MS). Upwards of 67% of patients present with MS-related CPS impairment, which is associated with poor everyday life outcomes. There are no FDA-approved pharmacological treatments for CPS impairment in MS. This landscape creates a critical public health and clinical crisis that underscores the importance of identifying efficacious approaches for managing CPS impairment in MS. We believe that aerobic exercise training represents a promising and powerful behavioral approach. This project involves a single-blind randomized controlled trial of 16-weeks of remotely-delivered and supported aerobic walking exercise training compared with an active control condition (remotely-delivered and supported stretching and toning activities) on CPS (assessed remotely) in 24 fully-ambulatory, but CPS-impaired persons with MS.

This pilot trial will be conducted in a fully-remote fashion, such that there are no required in-person visits to Kessler Foundation. Participants (N=24) will initially undertake baseline assessments of CPS remotely via a HIPAA-compliant virtual platform (i.e., Zoom for Healthcare). This assessment will also serve as a screen for ensuring impaired CPS. At this virtual study visit, participants further will undergo a neuropsychological test of verbal learning and complete questionnaires assessing physical activity and MS symptoms via computer (REDCap). Following baseline, participants will be randomly assigned into the remotely-delivered and supported aerobic walking exercise training intervention condition (n=12) or remotely-delivered and supported attention and social contact control condition (n=12) using concealment. Both conditions will be administered remotely over 16-weeks via telerehabilitation by a postdoctoral behavior coach during scheduled calls. Participants will undertake aerobic walking exercise training or stretching-and-toning in the home/community. The exercise training intervention involves aerobic walking exercise training that is monitored by a waist-worn FitBit and follows prescriptive guidelines for aerobic exercise for persons with MS. The control condition involves stretching-and-toning based on a manual published by the National Multiple Sclerosis Society. Both conditions further involve one-on-one coaching, action-planning via calendars, logs for self-monitoring, and newsletters based on Social Cognitive Theory. After the 16-week exercise/control period, participants will undergo remote assessments of CPS and verbal learning (administered by a treatment-blinded assessor) as well as completion of questionnaires assessing physical activity and MS symptoms via REDCap.

If successful, this RCT will provide preliminary data on the extent to which (a) remotely-delivered/supported aerobic walking ET results in significant CPS improvements in CPS-impaired persons with MS; and (b) the intervention results in increased physical activity relative to an active control in a cognitively-impaired cohort. These pilot data will be essential for supporting a large R01 application on a multi-site, effectiveness RCT in a nationwide sample of CPS-impaired persons with MS.

ELIGIBILITY:
1. MS Diagnosis: All participants must have a definite diagnosis of MS.
2. Most recent exacerbation: MS subjects will be free from exacerbations and not have acutely taken corticosteroids at least 30 days prior to enrollment.
3. Internet and email access: All participants must have Internet access on a device larger than a smartphone (i.e., full-size iPad, desktop, laptop) for standardizing the SDMT and CVLT-II, as well as for receiving the study conditions via Zoom for Healthcare, registering for Fitabase, and email for receiving updates on study processes and communication with the study staff.
4. Willingness to complete the measures and be randomized.
5. Physical activity status: All participants must be insufficiently physically active, based on a health contribution score of less than 14 units from the Godin Leisure-Time Exercise Questionnaire (GLTEQ). This is necessary for minimizing potential ceiling effects of the intervention condition on physical activity.
6. Ambulatory status: All participants will be able to walk without an assistive device, and have Patient-Determined Disease Steps (PDDS) scores between 0 and 2 for confirmation of being fully-ambulatory.
7. Fall risk: All participants will not have fallen due to MS in the past 6 months (i.e., low fall risk).
8. Age: All subjects will be between the ages of 18 and 65.
9. Psychiatric status: Participants will not have uncontrolled major depression disorder or a history of other significant psychiatric disorders (e.g., bipolar disorder I or II, schizophrenia).
10. Medications: Participants will not regularly be taking medications that can affect cognition, such as antipsychotics or benzodiazepines. Study staff will review self-reported medications to determine participant eligibility status.
11. Contraindications for ET: We will exclude all individuals with moderate or high risk for contraindications of possible injury or death when undertaking strenuous or maximal exercise using the Physical Activity Readiness Questionnaire (PAR-Q). During the initial phone contact with Ms. Wells, participants will verbally respond to the 7-items on the PAR-Q, and those individuals who report one or fewer YES or affirmative responses on the seven PAR-Q items will be considered at low risk and included for participation. All other individuals will be considered at moderate or high risk for starting a physical activity program and excluded from participation.
12. Severe cognitive impairment: Ms. Wells will administer the Telephone Interview for Cognitive Status (TICS-M) over the phone to ensure that all participants can adequately follow directions. In order to pass this inclusion criterion, participants must demonstrate TICS-M scores of 18 or higher. This is critical for ensuring that participants do not have severe cognitive impairment that might preclude the ability to adhere to the conditions, understand intervention content, and interact with the behavior coach.

If the prospective participant with MS passes the above screen, a second-level screening for CPS impairment will take place via Zoom:

a. CPS impairment: All participants will demonstrate impairment in CPS based on Symbol Digit Modalities Test (SDMT) scores at least 1 SD below the age-adjusted normative score for healthy controls.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2022-05-25 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Change in Cognitive Processing Speed | 16 weeks
  Cognitive processing speed will be measured using the Symbol Digit Modalities Test. The primary outcome measure is the total score.

SECONDARY OUTCOMES:
Change in Verbal Learning and Memory | 16 weeks
  Verbal learning and memory will be measured using the learning trials of the California Verbal Learning Test-II. The primary outcome measure is the total learning score.

CONTACTS AND LOCATIONS:
Locations (1):
- Kessler Foundation, West Orange, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No